CLINICAL TRIAL: NCT04217265
Title: Letrozole Pretreatment With Misoprostol for Induction of Abortion In First-Trimester Missed Miscarriage: A Randomized Controlled Trial
Brief Title: Letrozole Pretreatment With Misoprostol Versus Misoprostol Alone in Missed Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: letrozole
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 2 tablets of Letrozole 2.5 mg will be given as single daily doses, 5 mg per day for two days at home and the third dose will be given on admission to hospital on day 3 and will be followed by vaginal misoprostol 800 mcg every three hours up to maximum three doses.
  Interventions: Drug: Letrozole then misoprostol
- control group (Placebo Comparator): 2 tablets of placebo will be given as a single daily dose, for two days at home and will be admitted on day 3 and continue treatment with misoprostol 800 mcg every three hours up to maximum three doses
  Interventions: Drug: placebo then misoprostol

INTERVENTIONS:
Drug: Letrozole then misoprostol — total dose 5 mg per day for 3 days then Misoprosrol 800mcg will be given to all patients for induction of abortion
  Arms: study group
Drug: placebo then misoprostol — placebo tablets for 3 days then Misoprosrol 800mcg will be given to all patients for induction of abortion
  Arms: control group

SUMMARY:
This study compares the success rate of letrozole and misoprostol versus misoprostol alone for medical termination of first-trimester pregnancy.

DETAILED DESCRIPTION:
According to the American college of obstetricians and gynecologists (2005), medical abortion is an acceptable alternative for surgical procedures in pregnant women with gestational age of less than 49 days based on the last menstrual period

Oral or vaginal misoprostol causes complete abortion in almost 85% of cases within seven days before the 12th week

letrozole administration with misoprostol raises the rate of complete abortion

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 64 days gestation (<9 wks).
* Hemoglobin >10 g/dL.
* BMI between 18.5 kg/m2 and 25 kg/m2.
* Missed abortion.

Exclusion Criteria:

* Molar pregnancy.
* Fibroid uterus.
* Uterine anomalies.
* Coagulopathy.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.
* Scared uterus (previous myomectomy, cesarean section, hysterectomy and ruptured uterus).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-05 (Estimated); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
complete abortion rate | 9 hours
  Incidence of complete miscarriage
time from induction to abortion | 9 hours
  induction to abortion time interval

SECONDARY OUTCOMES:
Need for surgical evacuation of the products of conception | 9 hours
  how many women will undergo dilatation and curettage after failed medical induction of abortion

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University